CLINICAL TRIAL: NCT03391102
Title: Matão Preventing Stroke (MaPS): Stroke Register in City of Matão, Brazil
Brief Title: Matão Preventing Stroke (MaPS): a Stroke Register Study
Acronym: MaPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Neurológico de Pesquisa e Reabiitação, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: Cenp-Reab
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Stroke
Keywords: Epidemiology; Community-based study
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study

SUMMARY:
Stroke is one of the most important cause of mortality and disability in Brazil. The city of Matão, located in São Paulo state, with a population around 80.000 inhabitants, has conditions to develop a community-based stroke study, which can answer important questions regarding epidemiological data over the time.

Therefore, the purpose of this prospective community based study is to observe trends in stroke incidence, types and sub-types of stroke, risk factors, prognosis, 30 days and one year case-fatality during a follow-up of ten years.

This study offers the opportunity to conduct an epidemiological study of high quality which can obtain data to formulate public politics to reduce the social and economic impact of stroke in Brazil.

DETAILED DESCRIPTION:
Introduction

Community-based stroke studies can answer important questions regarding incidence, case fatality, recurrence, disability, assessment of risk factors and quality of stroke services.

Brazil had the highest age-adjusted stroke death rate of all Latin-American countries and the risk of premature death due to stroke is one of the highest in the world. Although, a decline in Brazilian stroke incidence and mortality has been observed in last years, stroke still has an important social burden in the country.

The purpose of this study is to observe trends in stroke incidence, types and sub-types of stroke, risk factors, prognosis, 30 days and one case-fatality during a follow-up of ten years.

Objectives

The objectives of this project is to analyze:

The incidence of first-ever-in-a-lifetime stroke and incidence of pathological types, subtypes, and rare causes Case fatalities Prognosis Early and long-term case-fatality rates Poststroke morbidity Disability and handicap pos-stroke Risk factors Complications after stroke Recurrent stroke Other vascular events Trends in stroke incidence

Subjects and Methods

Study Design A prospective population-based study is being performed since August, 1, 2015

Site of Investigation

Matão is a city located in São Paulo state, in the Brazilian southwest, 300 km northwest of the state capital. Matão population was 78.690 in 2015 and estimated population in 2025 is 80791 inhabitants. There is only 1 hospital in the city, which serves the whole city and 2 other small towns. This is a general secondary level public hospital, with 190 beds, including 18 beds in the intensive care unit and a radiology service with CT scan, the only one in the city. The emergency department attends to 5000 to 6000 people monthly; including emergency and urgency cases. The emergency department and intensive care unit take care of acute stroke patients according to a written protocol that includes hospitalization and a brain CT scan applied as soon as possible to all patients with suspected stroke.

Case Ascertainment All the physicians in the city are instructed to refer suspected acute stroke patients to the research team or to the hospital emergency department. The neurologists of the research team check all radiology records in suspected cases of stroke. The hospital admission and discharge lists are checked weekly, searching for any suspected case. All death certificates from the study period are checked monthly to search for stroke patients who died in their homes and are not been referred to the hospital.

Inclusion criteria All suspected stroke patients living in Matão at an address belonging to the city are included, regardless of age. The stroke criteria is rapidly developing clinical symptoms and/or signs of focal and at time global loss of cerebral function, with symptoms lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin. Only the first-ever-in-a-lifetime stroke is being included in the analysis.

Exclusion criteria Patients not living in Matão, who did not fulfill the clinical criteria for stroke, with CT scan findings incompatible with a clinical suspicion of stroke and with clinical evidence of a previous stroke event.

Follow-Up All included cases are being followed-up prospectively by the research team during the first, third, sixth, months and 1 year after the stroke event with hospital visits. Patients unable to attend the scheduled visits or who had moved to another city are being contacted by telephone.

Classifications and Definitions The subtypes of stroke are being classified as ischemic stroke and intracerebral hemorrhage on the basis of CT scan findings and subarachnoid hemorrhage on the basis of CT scan and cerebrospinal fluid findings. Ischemic stroke is subdivided into four subtypes according to the Oxfordshire Community Stroke Project classification. For prognosis, is considered independence in activities of daily living if patient reaches 100 points on the Barthel scale, independent gait if the patient reached 15 points in the mobility subsection of the Barthel scale, recurrent stroke if any new episode of focal cerebral dysfunction persisting 24 hours during the follow-up period.

Data Analysis The age- and sex-specific annual incidence of first-ever-stroke per 100 000 inhabitants it is being estimated according to the official system of the Brazilian Ministry of Health stratification and is presented as 10-year age bands as follows: younger than 45, 45 to 54, 55 to 64, 65 to 74, and 75 years or older. The incidence rate will be calculated as the number of cases divided by the population at risk in the specific age bands, according the respective year population. Inferential analyses will be performed by the 2-sided Fischer exact test, with the level of significance set at 5%.

Discussion

Population-based studies can identify all types and sub-types of stroke in a community. Studies including just data from hospitals, may not include mild stroke that are not hospitalized and also severe stroke that die at home and do not have hospitals admission.

Additionally, it is fundamental that this studies should be prospective and in a long follow-up. As diagnostic of stroke is basically clinical, prospective studies allow more specific methods to define the type of stroke, risk factors, impairments and handicaps over time.

The paucity of data regarding incidence on long follow-up and the distinct etiologies as cause of stroke are being responsible as the main causes of the high incidence and case fatality in the world. This study in Matão offers the opportunity to conduct an epidemiologic study of high quality, which will be able to obtain data to formulate public politics to reduce the social and economic impact of stroke in Brazil.

ELIGIBILITY:
Inclusion Criteria: All suspected stroke patients living in Matão at an address belonging to the city were included, regardless of age. The stroke criteria were those defined by the Word Health Organization: "rapidly developing clinical symptoms and/or signs of focal and at time global loss of cerebral function, with symptoms lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin" 12 Although every stroke was recorded, only the first-ever-in-a-lifetime stroke was included in the analysis.

Exclusion Criteria: Patients not living in Matão, who did not fulfill the clinical criteria for stroke, with CT or RMI scan findings incompatible with a clinical suspicion of stroke, and with clinical evidence of a previous stroke event.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population belongs to Matão, Brazil, São Paulo state, located 300 km northwest of the state capital. The number od inhabitants in 2014 was estimated in 78.910 and in 2025, 80.791 habitants, with no difference in sex distribution.
  The economy is mainly based on agricultural and industrial activities and on general services. Ethnicity is diverse, but most people are of white ethnicity, descendants of European immigrants. The population is urban and stable, with a low rate of interurban migration. Approximately 95% of all dwellings have piped water, a sewage network, and electricity.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Annual incidence of first-ever-stroke per 100 000 inhabitants | 1 year
  Number of first-ever stroke divided by the population at risk.

CONTACTS AND LOCATIONS:
Overall Officials: Cesar Minelli, PhD,, Principal Investigator — Hospital Carlos Fernando Malzoni
Locations (1):
- Hospital Carlos Fernando Malzoni, Matão, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data regarding demography and prognosis can be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become avaliable on July, 2018
Access Criteria: Researches interested in stroke epidemiology

REFERENCES:
- [Result] Sudlow CL, Warlow CP. Comparing stroke incidence worldwide: what makes studies comparable? Stroke. 1996 Mar;27(3):550-8. doi: 10.1161/01.str.27.3.550. PMID 8610328
- [Result] Ribeiro AL, Duncan BB, Brant LC, Lotufo PA, Mill JG, Barreto SM. Cardiovascular Health in Brazil: Trends and Perspectives. Circulation. 2016 Jan 26;133(4):422-33. doi: 10.1161/CIRCULATIONAHA.114.008727. PMID 26811272
- [Result] Cabral NL, Cougo-Pinto PT, Magalhaes PS, Longo AL, Moro CH, Amaral CH, Costa G, Reis FI, Goncalves AR, Nagel V, Pontes-Neto OM. Trends of Stroke Incidence from 1995 to 2013 in Joinville, Brazil. Neuroepidemiology. 2016;46(4):273-81. doi: 10.1159/000445060. Epub 2016 Apr 12. PMID 27064414
- [Result] Bamford J, Sandercock P, Dennis M, Warlow C, Jones L, McPherson K, Vessey M, Fowler G, Molyneux A, Hughes T, et al. A prospective study of acute cerebrovascular disease in the community: the Oxfordshire Community Stroke Project 1981-86. 1. Methodology, demography and incident cases of first-ever stroke. J Neurol Neurosurg Psychiatry. 1988 Nov;51(11):1373-80. doi: 10.1136/jnnp.51.11.1373. PMID 3266234
- See also: population stratification by age bands — http://www.ibge.gov.br/apps/populacao/projecao/